CLINICAL TRIAL: NCT04137770
Title: Application of the ICE-T Postoperative Multimodal Pain Regimen to Laparoscopic Hysterectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment, change of OR policies due to COVID
Sponsor: Mercy Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-002
Record Dates: First submitted 2019-10-18; First posted 2019-10-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): Patients will receive routine post-operative analgesics
- intervention (Experimental): Patients will receive routine post-operative analgesics plus scheduled ketorolac and surgical site ice packs
  Interventions: Other: Ice pack and ketorolac

INTERVENTIONS:
Other: Ice pack and ketorolac — Scheduled IV ketorolac will be administered and ice packs will be applied to the surgical site
  Arms: intervention

SUMMARY:
This is a randomized controlled trial evaluating whether application of ice packs and scheduled ketorolac to the surgical site after laparoscopic hysterectomy reduces need for narcotic medications.

DETAILED DESCRIPTION:
Patients who undergo laparoscopic hysterectomy and chose to participate in the study will be randomized to either receive the standard post-surgical analgesic protocol (control group) or the standard post-surgical analgesic protocol plus scheduled ketorolac and surgical site ice packs. Usage of narcotic analgesics for breakthrough pain will be monitored and compared between cohorts. All care received by test subjects will be standard of care, with the only difference being the use of ice packs and scheduled ketorolac.

ELIGIBILITY:
Inclusion Criteria:

Females, 18-65 years old at time of new patient evaluation, Planned laparoscopic hysterectomy only or hysterectomy with or without unilateral or bilateral oophorectomy or salpingo-oophorectomy by Dr. Corey Wagner, Uterus with expected size greater than 250 grams as determined by bimanual exam or standard of care ultrasound obtained prior to or as part of new patient evaluation

Exclusion Criteria:

Diagnosed or suspected endometriosis, Diagnosis of malignant carcinoma of the uterus, ovaries, or fallopian tubes, Diagnosis of severe renal disease (as determined by a GFR of less than 45), Known nonsteroidal anti-inflammatory drug (NSAID) intolerance, History of myocardial infarction, stroke or other cardiovascular disease, Known hypersensitivity or allergic reactions to Acetaminophen, Toradol, Ibuprofen, other NSAIDs, Aspirin or Roxicodone, Previous diagnosis of liver disease or hepatitis, Unable to take Tylenol (acetaminophen), Pre-existing narcotic drug regimens or opioid use disorders, Known diagnosis of or history of peptic ulcer disease, gastrointestinal bleeding or perforation, Known or suspected gastrointestinal obstruction including paralytic ileus, Diagnosis of severe bronchial asthma, Known diagnosis or history of cerebrovascular bleeding, Known bleeding disorder or coagulopathy based on patient history unless excluded by appropriate hematological examination, Daily prescription NSAID use, Adults unable to consent, Pregnancy as determined by urine or serum pregnancy test obtained in women of child-bearing age, Prisoners, Individuals who do not read and understand English

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Opioid analgesic usage in the 24 hours immediate post-operative period | 24 hours
  Opioid analgesic usage in the 24 hours immediately post-operative as measured in Morphine Milligram Equivalents

SECONDARY OUTCOMES:
Opioid analgesic usage for 6 weeks post-operative | 6 weeks
  Opioid analgesic usage for 6 weeks post-operative as measured in Morphine Milligram Equivalents
Pain scores in the 24 hours immediate post-operative period | 24 hours
  Pain scores (on a scale of 1-10, 10 being worse pain) as documented by the floor nurse in the patient's chart in the 24 hours immediate post-operative period

CONTACTS AND LOCATIONS:
Overall Officials: Corey A Wagner, MD, Principal Investigator — Mercy St. Louis
Locations (1):
- Mercy Hospital St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No